CLINICAL TRIAL: NCT01379040
Title: Detection of Pulmonary Colonization in Cystic Fibrosis Patients
Brief Title: Volatile Organic Compounds in Cystic Fibrosis
Acronym: VOCCF
Status: Completed | Type: Observational
Sponsor: Landon Pediatric Foundation (Other)
Responsible Party: Principal Investigator, Chris Landon, Principal Investigator, Landon Pediatric Foundation
Other Study IDs: CF1
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Cystic Fibrosis; Pseudomonas Aeruginosa
Keywords: Cystic Fibrosis; Pseudomonas aeruginosa; Volatile Organic Compounds; Electronic nose; Gas Chromatography
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cystic Fibrosis Patients: Patients with Cystic Fibrosis, some having Pseudomonas aeruginosa, some not.
  Interventions: Other: Cystic Fibrosis patients
- Control: Healthy volunteers

INTERVENTIONS:
Other: Cystic Fibrosis patients
  Groups: Cystic Fibrosis Patients

SUMMARY:
This experiment is designed to test the effectiveness of a new electronic nose device, which allows a non-invasive breath test for markers of lower respiratory tract infection, which may predict the probability of bacterial organisms in the lower respiratory tract. It consists of:

* A breath collection apparatus for collection of volatile organic compounds in breath onto a sorbent trap and Tedlar bag, as well as for the collection of a separate sample of room air.
* Analysis of the volatile organic compounds in breath and room air by short acoustic wave/gas chromatography.
* Interpretation of the volatile organic compounds with a proprietary algorithm in order to predict the probability of lower respiratory tract colonization and infection.

This study will test the hypothesis that the investigators can identify the presence of Pseudomonas aeruginosa by sampling the "head space" above culture media of sputum provided by patients with cystic fibrosis. This study will test the additional hypothesis that the investigators can identify the presence of Pseudomonas aeruginosa by sampling exhaled breath from the patient providing the sputum.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Cystic Fibrosis
* Must be able to give breath and sputum samples

Exclusion Criteria:

* Heavy smoker
* Inability to regularly give breath and sputum samples
* History of additional pulmonary disease

Ages: 1 Year to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients will be selected from Dr. Landon's primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Bacterial Identification | six months
  Patient's provided breath samples and sputum for culture. Bacterial identification by indices was achieved

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Diagnostic Center, Ventura, California, United States

REFERENCES:
- [Result] http://www.beehive.co.jp/est/samplePDF/CysticFibrosis.pdf